CLINICAL TRIAL: NCT01146470
Title: A Single-Center, Double-blind, Random, Parallel Controlled Study
Brief Title: The Influence of Red Grape Cells on Blood Pressure Vascular Function in People With Hypertension
Acronym: RGC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Fruitura Bioscience Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TASMC-10-NV-0176-CTIL; RGC
Record Dates: First submitted 2010-06-16; First posted 2010-06-17 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2010-06

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- RGC 200 mg (Experimental)
  Interventions: Dietary Supplement: RGC
- RGC 400 mg (Experimental)
  Interventions: Dietary Supplement: RGC
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: RGC — dosage of Red Grape Cells once a day, during 3 months
  Arms: RGC 200 mg; RGC 400 mg
Dietary Supplement: Placebo — dosage of Placebo once a day, during 3 months
  Arms: Placebo

SUMMARY:
The study hypothesis is that 3 Months Daily Supplementation of RGC will effect blood pressure and vascular function.

This will be a single-center, double-blind, random, parallel controlled Study. Study population will include 60 subjects, who will be divided randomly into three groups. The first group will get RGC 200mg, the second group will get RGC 400mg, and the third group will get 200mg placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age 35-70
* BMI < 40.0 kg/m2
* Blood pressure: SYS. ≤154 mmHg, DIA. ≤93 mmHg.

Exclusion Criteria:

* Breastfeeding or pregnancy.
* Milk allergy - the substance may contain traces of milk protein (casein).
* Taking anti-hypertensive medications.
* Taking antioxidant food supplements, excluding probiotic agents and fibers (taken for less than two weeks before beginning the study).
* Subjects suffering from any of the following conditions: cardiovascular disorders, renal disorders, intestinal disorders, hepatic disease, malignant or autoimmune diseases or other metabolic diseases.
* A subject whose baseline blood tests indicate abnormalities in hepatic or renal function, thyroid function or blood count.
* Unusual eating habits.
* The subject is in the process of active weight loss / gain.
* Addiction to drugs / alcohol.
* Medically documented psychiatric problems or neurological disorders.
* Smokers. (Subjects who quit smoking more than two years ago may be included in the study).
* Systolic blood pressure above 154 mmHg.
* Diastolic blood pressure above 93 mmHg.
* Taking phosphodiesterase 5 inhibitors for the treatment of erectile dysfunction (Viagra, Cialis, etc.).

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-07; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
To investigate the influence of RGC on blood pressure and vascular function. | 3 months of treatment

SECONDARY OUTCOMES:
The change in oxidative stress parameters | 3 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Nachum Vaisman, Professor, Principal Investigator — Tel-Aviv Sourasky Medical Center, Israel
Locations (1):
- Tel Aviv Medical Center, Tel Aviv, Israel